CLINICAL TRIAL: NCT01584934
Title: The Effect of Sodium Oxybate in Patients With Chronic Fatigue Syndrome.
Brief Title: Sodium Oxybate in Patients With Chronic Fatigue Syndrome.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: incompatibilities over intellectual property
Sponsor: University Hospital, Ghent (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012/197; 2011-006336-23 (EudraCT Number)
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Chronic Fatigue Syndrome
Keywords: fatigue; sleep quality; Chronic, disabling, unexplained fatigue with at least 4 minor criteria for CFS, according to the 1994 Fukuda case definition
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue; Sleep Initiation and Maintenance Disorders; Bronchiolitis Obliterans Syndrome | interventions — Sodium Oxybate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium oxybate (Experimental): Patient group receives sodium oxybate as treatment.
  Interventions: Drug: Sodium oxybate
- Placebo (Placebo Comparator): Patient group receives placebo as treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium oxybate — Treatment is started and continued for 6 weeks at patient's home. Patients receive 3g/night during the first week, and 4,5 g/night during the second week. After the second week, patients have their dose increased to 6 g/night during 6 weeks. A washout period of 4 weeks is installed to withdraw from treatment. Patients receive 4,5 g/night for 1 week, followed by 3g/night for 1 week. The next 2 weeks, patients are not treated.
  Arms: Sodium oxybate
Drug: Placebo — Placebo treatment is started and continued for 6 weeks at patient's home. Patients receive 3 g/night during the first week and 4.5 g/night during the second week. After the second week, patients have their dose increased to 6 g/night during 6 weeks. A washout period of 4 weeks is installed to withdraw from treatment. Patients receive 4.5 g/night for 1 week, followed by 3 g/night for 1 week. The next 2 weeks, patients are not treated.
  Arms: Placebo

SUMMARY:
Chronic fatigue syndrome (CFS) is a disabling, unexplained disorder characterized by physical and mental exhaustion. Complaints of disturbed and unrefreshing sleep are very common in CFS patients, however, the relationship between (disturbed) sleep quality and fatigue is still not fully elucidated. To evaluate the effect of sodium oxybate on fatigue and to explore the interdependence of sleep quality and fatigue in CFS, a double blind, randomized, placebo controlled cross-over trial with sodium oxybate is carried out in CFS patients.

The aim of this study is to address the issue of the effect of sodium oxybate on fatigue as a presenting symptom in chronic fatigue (CF) and CFS patients, in the absence of underlying medical or psychiatric illness. The answer to this question may shed further light on the enigmatic relationship between sleep and fatigue. We also want to investigate the effect of sodium oxybate on sleepiness and general health in the same target population.

Zero-hypothesis: there is no effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from chronic, disabling, unexplained fatigue with at least 4 minor criteria for CFS, according to the 1994 Fukuda case definition;
* Negatively screened for fibromyalgia syndrome(FMS) according to the American College of Rheumatology (ACR) classification criteria;
* 18 years or older;
* 65 years or less;
* Female patient of childbearing potential (premenopausal female biologically capable of becoming pregnant) has a confirmed negative pregnancy test at the start of the trial and has to employ an acceptable method of birth control (double barrier method of contraception);
* Written, signed and dated informed consent must be obtained from each patient;
* Patient able to understand and follow the requirements of the study
* Willing to abstain from taking any medication or treatment prohibited in the protocol

Exclusion Criteria:

* FMS;
* Presence of an inflammatory rheumatic disease or a painful disorder other than FMS;
* Fatigue that is explained by medical or psychiatric causes;
* Older than 65 or younger than 18 years of age;
* Apnea/hypopnea index (AHI) > or equal to 15 on polysomnography (PSG) (exempted if receiving continuous positive airway pressure CPAP and shown good compliance)
* Deficiency in succinic semialdehyde dehydrogenase;
* Porphyria;
* Breathing or lung problems;
* Unsufficiently controlled hypertension (high blood pressure: > 140/90 mmHg);
* Heart failure;
* Liver or kidney problems (serum creatinine level > 2,0 mg/dl);
* Presence of a seizure disorder or epilepsy;
* Sodium oxybate treatment in the past;
* Primary history of substance abuse (including abuse of alcohol);
* Inability to withdraw from psychoactive drugs;
* Current use of sedative (benzodiazepine and non-benzodiazepine GABA-ergic agonists), opioids or antidepressant medication or a drug-free interval of less than 4 weeks;
* Female patient who is pregnant, lactating or has a positive pregnancy test result.
* Occupation that requires night-shift work;
* Willing to abstain from using alcohol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Measurement of the effect of sodium oxybate on fatigue with questionnaires. | before treatment (baseline evaluation)
  Questionnaires: Visual Analog Scale (VAS), fatigue severity scale (FSS) and checklist individual strength (CIS).
Measurement of the effect of sodium oxybate on fatigue with questionnaires. | after 42 days of first treatment
  Questionnaires: Visual Analog Scale (VAS), fatigue severity scale (FSS) and checklist individual strength (CIS).
Measurement of the effect of sodium oxybate on fatigue with questionnaires. | after 42 days of second treatment (113 days after baseline)
  Questionnaires: Visual Analog Scale (VAS), fatigue severity scale (FSS) and checklist individual strength (CIS).

SECONDARY OUTCOMES:
Effect of sodium oxybate on sleepiness. | before treatment (baseline evaluation)
  Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), Medical Outcomes Study 36-item Short Form health survey (MOS SF-36), Visual Analogue Scale for Pain (VAS-P), Multidimensional Pain Inventory (MPI), Polysomnography, multiple sleep latency test.
Effect of sodium oxybate on sleepiness | after 42 days of first treatment
  Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), Medical Outcomes Study 36-item Short Form health survey (MOS SF-36), Visual Analogue Scale for Pain (VAS-P), Multidimensional Pain Inventory (MPI), Polysomnography, multiple sleep latency test.
Effect of sodium oxybate on sleepiness. | after 42 days of second treatment (113 days after baseline)
  Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), Medical Outcomes Study 36-item Short Form health survey (MOS SF-36), Visual Analogue Scale for Pain (VAS-P), Multidimensional Pain Inventory (MPI), Polysomnography, multiple sleep latency test.
Effect of sodium oxybate on sleep quality. | before treatment (baseline evaluation)
  Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), Medical Outcomes Study 36-item Short Form health survey (MOS SF-36), Visual Analogue Scale for Pain (VAS-P), Multidimensional Pain Inventory (MPI), Polysomnography, multiple sleep latency test.
Effect of sodium oxybate on sleep quality. | 42 days after first treatment
  Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), Medical Outcomes Study 36-item Short Form health survey (MOS SF-36), Visual Analogue Scale for Pain (VAS-P), Multidimensional Pain Inventory (MPI), Polysomnography, multiple sleep latency test.
Effect of sodium oxybate on sleep quality. | 42 days after second treatment (113 days after baseline)
  Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), Medical Outcomes Study 36-item Short Form health survey (MOS SF-36), Visual Analogue Scale for Pain (VAS-P), Multidimensional Pain Inventory (MPI), Polysomnography, multiple sleep latency test.
Effect of sodium oxybate on general health. | before treatment (baseline evaluation)
  Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), Medical Outcomes Study 36-item Short Form health survey (MOS SF-36), Visual Analogue Scale for Pain (VAS-P), Multidimensional Pain Inventory (MPI), Polysomnography, multiple sleep latency test.
Effect of sodium oxybate on general health. | 42 days after first treatment
  Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), Medical Outcomes Study 36-item Short Form health survey (MOS SF-36), Visual Analogue Scale for Pain (VAS-P), Multidimensional Pain Inventory (MPI), Polysomnography, multiple sleep latency test.
Effect of sodium oxybate on general health. | 42 days after second treatment (113 days after baseline)
  Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), Medical Outcomes Study 36-item Short Form health survey (MOS SF-36), Visual Analogue Scale for Pain (VAS-P), Multidimensional Pain Inventory (MPI), Polysomnography, multiple sleep latency test.
Effect of sodium oxybate on pain. | before treatment (baseline evaluation)
  Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), Medical Outcomes Study 36-item Short Form health survey (MOS SF-36), Visual Analogue Scale for Pain (VAS-P), Multidimensional Pain Inventory (MPI), Polysomnography, multiple sleep latency test.
Effect of sodium oxybate on pain. | 42 days after first treatment
  Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), Medical Outcomes Study 36-item Short Form health survey (MOS SF-36), Visual Analogue Scale for Pain (VAS-P), Multidimensional Pain Inventory (MPI), Polysomnography, multiple sleep latency test.
Effect of sodium oxybate on pain. | 42 days after second treatment (113 days after baseline)
  Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI), Medical Outcomes Study 36-item Short Form health survey (MOS SF-36), Visual Analogue Scale for Pain (VAS-P), Multidimensional Pain Inventory (MPI), Polysomnography, multiple sleep latency test.

CONTACTS AND LOCATIONS:
Overall Officials: An Mariman, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be